CLINICAL TRIAL: NCT00019591
Title: A Phase I/II Trial of Vaccination With Mutant Ras Peptide-Pulsed Dendritic Cells in the Treatment of HLA A2.1 Positive Patients With Colorectal Cancer
Brief Title: Vaccine Therapy With or Without Interleukin-2 in Treating Patients With Locally Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066874; NCI-99-C-0023L; NCI-T98-0034; NCT00001794 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-11

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — aldesleukin; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: ras peptide cancer vaccine
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response that will kill cancer cells. Combining vaccine therapy with interleukin-2 may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy with or without interleukin-2 in treating patients who have locally advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of immunologic response in patients with locally advanced or metastatic colorectal cancer treated with ras peptide-pulsed dendritic cell vaccine with or without interleukin-2.
* Determine the tumor response and survival time in patients with metastatic colorectal cancer treated with vaccine plus interleukin-2.
* Determine the time to progression in patients with locally advanced colorectal cancer treated with adjuvant vaccine.

OUTLINE: Patients are assigned to 1 of 2 treatment groups according to extent of disease. Patients with prior locally advanced disease are assigned to treatment group A, while those with metastatic disease are assigned to treatment group B.

* Group A: Patients are vaccinated against influenza on day -6. Patients undergo collection of peripheral blood mononuclear cells (PBMC) on day -4. The PBMC are cultured with sargramostim (GM-CSF) and interleukin-4 for 5 days and CD40 ligand for 24 hours and then pulsed for 2 hours with the appropriate peptide to form a vaccine. Patients receive ras peptide-pulsed dendritic cell vaccine IV over 5 minutes on days 1, 15, 29, 43, and 57.
* Group B: Patients undergo collection of PBMC and receive vaccination as in group A. Patients also receive interleukin-2 subcutaneously on days 2-6 and 9-13.

Treatment in both groups repeats every 2 weeks for up to 5 vaccinations in the absence of disease progression or unacceptable toxicity.

Patients are followed on days 75, 90, 120, and 365.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced or metastatic colorectal cancer
* Metastatic disease must be radiologically proven
* HLA-A2-1 positive
* Locally advanced disease must have had prior resection or incomplete resection with poor prognosis
* Locally advanced disease includes:

  * Stage III or IV colon cancer (T4 or any T, N2-3, M0)
  * Stage III or IV rectal cancer (T4 or T3, N1-3)
  * Resectable or unresectable T4 disease after radiotherapy, chemotherapy, and/or surgery
  * Absence of measurable disease but more than a 50% chance of recurrence
* Completely resected or locally advanced disease may have had conventional therapy completed within 1-12 months (surgery alone, with or without adjuvant chemotherapy and/or radiotherapy) prior to study entry
* Metastatic disease patients must have bidimensionally measurable disease

  * Bone lesions with well-demarcated borders allowed
  * Lesions seen only on bone scan, pleural effusions, ascites, and changes in carcinoembryonic antigen are not considered measurable disease

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Lymphocyte count at least 470/mm^3
* Granulocyte count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL*
* SGOT no greater than 4 times upper limit of normal (ULN) (2.5 times ULN for adjuvant patients)*
* Albumin at least 3 g/dL
* No active viral hepatitis
* No evidence of chronic infection due to hepatitis C
* Hepatitis B surface antigen negative NOTE: *Unless due to metastatic disease

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No history of cardiac failure, significant arrhythmias, or coronary artery disease (metastatic disease patients only)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No prior malignancy with a 50% chance of recurrence within 5 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No medical or psychiatric condition that would preclude compliance
* No serious medical condition that would preclude apheresis
* No serious infection
* No uncontrolled thyroid disease (metastatic disease patients only)
* Patients with an allergy to eggs are allowed but are not vaccinated against influenza during study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunologic therapy directed at the cellular immune system

Chemotherapy:

* See Disease Characteristics
* Prior chemotherapy for metastatic disease allowed
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy or anticipated need for chemotherapy for 2 months after vaccinations

Endocrine therapy:

* At least 4 weeks since prior supraphysiologic steroid therapy

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy for metastatic disease allowed
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Prior surgery for metastatic disease allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Response rate every 3 months for up to a year after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: John E. Janik, MD, Study Chair — NCI - Metabolism Branch;MET
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee